CLINICAL TRIAL: NCT04198662
Title: Intercostal Cryoneurolysis Following Traumatic Rib Fractures
Brief Title: Rib Fracture Analgesia Using Cryoanalgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rib Fracture & Spirometry/Cryo
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Rib Fracture(s)
MeSH Terms: interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-masked, sham-controlled, parallel design, clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization lists will be created by the UC San Diego Investigational Drug Service which will create the sealed, opaque randomization envelopes with treatment group assignments. The treating investigators doing the procedures will be the only other individuals aware of the treatment group assignments. The Investigational Drug Service will not provide the treatment group assignments to the investigators until the completion of data collection for all subjects; and will only provide "Treatment A" vs "Treatment B" assignments for the initial statistical analysis. Only at the completion of statistical analysis will each treatment be revealed to the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis and placebo intercostal nerve block (Active Comparator): Active cryoneurolysis: 3 mL of normal SALINE will be injected into the muscle superficial to the nerve followed by an ACTIVE cryoneurolysis procedure using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods.
  Interventions: Device: Cryoneurolysis with a Painblocker (Epimed International, Farmers Branch, Texas); Drug: Placebo intercostal nerve block with normal saline
- Sham cryoneurolysis and active intercostal nerve block (Sham Comparator): Sham cryoneurolysis: 3 mL of ropivacaine 0.5% (with epinephrine) will be injected perineurally to provide the intercostal nerve block followed by a SHAM cryoneurolysis procedure with a probe that vents the nitrous oxide prior to reaching the probe tip using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods.
  Interventions: Drug: Intercostal nerve block ropivacaine with epinephrine; Device: Sham cryoneurolysis with a Painblocker

INTERVENTIONS:
Device: Cryoneurolysis with a Painblocker (Epimed International, Farmers Branch, Texas) — The cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Arms: Cryoneurolysis and placebo intercostal nerve block
Drug: Intercostal nerve block ropivacaine with epinephrine — 3 mL of ropivacaine 0.5% (with epinephrine) will be injected perineurally to provide the intercostal nerve block(s)
  Arms: Sham cryoneurolysis and active intercostal nerve block
Device: Sham cryoneurolysis with a Painblocker — The cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods. For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change.
  Arms: Sham cryoneurolysis and active intercostal nerve block
Drug: Placebo intercostal nerve block with normal saline — 3 mL of normal saline will be injected perineurally to provide placebo intercostal nerve blocks
  Arms: Cryoneurolysis and placebo intercostal nerve block

SUMMARY:
Rib fractures are one of the most common injuries in trauma patients. These fractures are associated with significant pain as well as decreased ability to inspire deeply or cough to clear secretions, which together lead to pulmonary complications and a high degree of morbidity and mortality. Peripheral nerve blocks as well as epidural blocks have been used with success to improve pain control in rib fracture patients and have been associated with decreased pulmonary complications and improved outcomes. However, a single-injection nerve block lasts less than 24 hours; and, even a continuous nerve block is generally limited to 3-4 days. The pain from rib fractures usually persists for multiple weeks or months. In contrast to local anesthetic-induced nerve blocks, a prolonged block lasting a few weeks/months may be provided by freezing the nerve using a process called "cryoneurolysis". The goal of this multicenter, randomized, double-masked, sham-controlled, parallel-arm study is to evaluate the potential of cryoanalgesia to decrease pain and improve pulmonary mechanics in patients with rib fractures.

DETAILED DESCRIPTION:
The ultimate objective of the proposed line of research is to determine if cryoanalgesia is an effective treatment for pain associated with rib fractures; and, if this analgesic modality improves pulmonary mechanics measured with incentive spirometry.

Specific Aim 1: To determine if, compared with current and customary analgesia for rib fracture(s), intercostal nerve cryoneurolysis improves maximum inspiratory volume.

Hypothesis 1a: The maximum inspired volume will be significantly increased on the day following the procedure [primary endpoint] as well as at other time points following the procedure [secondary end points] with intercostal cryoanalgesia as compared single-injection local anesthetic-based intercostal nerve blocks [measured with an incentive spirometer].

Hypothesis 1b: The maximum inspired volume as a percentage of the baseline will be significantly increased on the day following the procedure [secondary endpoint of greatest interest], as well as at other time points following the procedure [secondary end points] with intercostal cryoanalgesia as compared with single-injection local anesthetic-based intercostal nerve blocks [measured with an incentive spirometer].

Specific Aim 2: To determine if, compared with current and customary analgesia, intercostal nerve cryoneurolysis decreases the pain associated with rib fracture(s).

Hypothesis 2a: The severity of rib fracture pain at rest will be significantly decreased within the 12 months following the procedure with intercostal cryoneurolysis as compared with subjects receiving single-injection local anesthetic-based intercostal nerve blocks [measured using the Numeric Rating Scale for pain].

Hypothesis 2b: The severity of rib fracture pain when using the spirometer or coughing will be significantly decreased within the 12 months following the procedure with intercostal cryoneurolysis as compared with subjects receiving single-injection local anesthetic-based intercostal nerve blocks [measured using the Numeric Rating Scale for pain].

Hypothesis 2c: The incidence of chronic pain will be significantly decreased 6 and 12 months following a rib fracture with intercostal cryoeurolysis as compared with subjects receiving single-injection local anesthetic-based intercostal nerve blocks [measured using the Numeric Rating Scale for pain].

Hypothesis 2d: The severity of chronic pain will be significantly decreased 6 and 12 months following a rib fracture with intercostal cryoneurolysis as compared with subjects receiving single-injection local anesthetic-based intercostal nerve blocks [measured using the Numeric Rating Scale for pain].

Study Overview Day 0 Baseline pain levels and spirometry Subjects randomized and cryoneurolysis/sham procedure administered Post-block pain levels and spirometry repeated

Days 1, 2, 7 Pain levels, opioid consumption, sleep disturbances due to pain, and incentive spirometry values collected [as well as the day of discharge]

Months 0.5, 1, 1.5 , 2, 3, 6, and 12 Pain levels, opioid consumption, sleep disturbances due to pain, and pain interference collected [and incentive spirometry if subject has spirometer available]

Subjects will be individuals who present to one of the UCSD hospitals with rib fracture(s) and significant pain. All will be following the same protocol and the subjects from all institutions will be combined for the analysis.

Treatment group assignment (randomization). Subjects will be allocated to one of two possible treatments stratified by unilateral vs. bilateral fractures:

1. active cryoneurolysis (sham local anesthetic intercostal blocks)
2. sham cryoneurolysis (active local anesthetic intercostal blocks)

Computer-generated randomization lists created by the UC San Diego Investigational Drug Service will be used to create sealed, opaque randomization envelopes with the treatment group assignment enclosed in each envelope labeled with the randomization number. The lists will be kept by the Investigational Drug Service and not provided to the investigators until completion of data collection (1 year following enrollment of the final subject).

The specific intercostal nerves targeted will depend on the injury site. The treatment sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Using the optimal ultrasound transducer for the specific anatomic location and subject anatomy (linear vs curvilinear array), the target nerves will be identified in a transverse cross-sectional (short axis) view. The intercostal nerve of each fractured rib as well as the level above and below will be treated with the protocol below:

Intercostal nerve block procedure: The target nerve will be visualized with ultrasound. Local anesthetic (1% lidocaine) will be used to infiltrate the skin and underlying muscle at each entry point. A 20 g Tuohy needle will be introduced through the skin wheel and along the anesthetized muscle tract. For subjects randomized to active cryo, 3 mL of normal saline will be injected into the muscle superficial to the nerve; and for subjects randomized to sham cryo, 3 mL of ropivacaine 0.5% (with epinephrine) will be injected perineurally to provide the intercostal nerve block.

Cryoneurolysis procedure: Cryoneurolysis probes are available for a console neurolysis device (PainBlocker, Epimed, Farmers Branch, Texas) that either (1) pass nitrous oxide to the tip inducing freezing temperatures; or, (2) vent the nitrous oxide at the base of the probe so that no gas reaches the probe tip, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected. An angiocatheter/introducer will be inserted beneath the ultrasound transducer and directed until the probe tip is immediately adjacent to the target nerve. The angiocatheter needle will be removed, leaving the angiocatheter through which the appropriate Epimed probe will be inserted until it is adjacent to the target nerve. The cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation (active or sham) separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis. For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change.

The process will be repeated with the same treatment probe for any additional nerves (e.g., all nerves will receive either active cryoneurolysis or sham/placebo, and not a mix of the two possible treatments).

Statistical Analysis: The primary endpoint is the maximum inspired volume measured by incentive spirometry the day following treatment. There is no accepted minimal clinically-relevant change in incentive spirometry volume. However, the median (IQR) of inspired volume for patients with rib fracture(s) is 1250 (750-1750) mL; and, ISV<1000 mL is associated with an increased risk of acute respiratory failure. The investigators will therefore use the difference between 1250 and 1000 (250 mL) as the minimal clinically-relevant difference. However, there is high variability in the reported increase in inspired volume with various regional analgesic interventions such as continuous intercostal nerve blocks and serratus plane blocks, and the investigators will therefore increase our enrollment to account for an unpredicted increase in variability or non-normal data distribution.

But, assuming a normal distribution, the interquartile range is approximately 1.35 standard deviations (SDs). Therefore an interquartile range of 250-50 = 200 mL (Hernandez et al. 2019) corresponds to, approximately, an SD of 200/1.35 = 148 mL. Assuming this SD of 148 mL, a sample size of n=7 per group provides 80% power to detect a group difference of d=250 mL per group with two sided Type 1 Error 5%. To allow for a larger-than-anticipated SD, we will enroll 10 subjects per group with an evaluable primary outcome measure (n=20 for both groups combined). Accounting for drop-outs, we request a maximum enrollment of 30 subjects.

Continuous data will be summarized with mean, SDs, medians, quartiles, and ranges; and displayed with box-and-whisker plots by group and in aggregate. Key baseline characteristics will be tested between groups using two-sample t-tests, and summarized with Cohen's D, for continuous measures; and Fisher's Exact test for categorical variables. The primary outcome is maximum incentive spirometry volume (ISV) measured in mL on POD 1. The group difference will be tested using Welch's two-sample test. Secondary outcomes will also be tested with the two-sample t-test. No multiplicity adjustments will be applied for these secondary outcomes. The Wilcoxon signed-rank test will be used as a sensitivity analysis. Secondary analyses will include a Mixed Model of Repeated Measures with fixed-effects for time, time-by-group, unilateral vs bilateral, and the number of fractures. The model will treat time as a categorical variable and will assume a compound symmetric correlation and heterogeneous variance with respect to time. The estimated mean difference between groups at the final scheduled timepoint will be the parameter of interest and will be tested using Kenward-Roger degrees of freedom. Outcomes only measured at baseline and a single follow-up timepoint will be analyses with Analysis of Covariance (ANCOVA). The dependent variable will be change from baseline, and covariates will include group, baseline outcome, unilateral vs bilateral, and the number of fractures. Missing data is not expected due to the short follow-up in this study. However, if missing data issues arise, the investigators will use multiple imputation which is robust to covariate-dependent Missing at Random, and tipping point analyses under various Missing Not at Random assumptions.

The Investigational Drug Pharmacists and investigators doing the study procedures will be the only individuals aware of the treatment group assignments. The Investigational Drug Service will not provide the treatment group assignments to the investigators until the completion of data collection for all subjects; and will only provide "Treatment A" vs "Treatment B" assignments for the initial statistical analysis. Only at the completion of statistical analysis will each treatment be revealed to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of at least 18 years of age
* having a total of 1-6 rib fractures at least 3 cm distal to the costo-transverse joint sustained within the previous 3 days (bilateral fractures are acceptable, but the total of the two sides combined must not exceed 6 fractures)
* regional anesthetic requested by the admitting service
* accepting of a cryoneurolysis procedure

Exclusion Criteria:

* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks
* pregnancy
* incarceration
* inability to communicate with the investigators
* morbid obesity (body mass index > 40 kg/m2)
* possessing any contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria and Reynaud's Syndrome
* any patient unable to correctly perform incentive spirometry as this is the primary outcome measure
* any patient with any degree of decreased mental capacity as determined by the surgical service
* any reason an investigator believes study participation would not be in the best interest of the potential subject
* flail chest
* chest tube
* fracture of the 1st rib on either side
* any moderate or severe pain (NRS>3) unrelated to the rib fracture(s), as best determined by the patient and investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (19) | 57 (14) | 52 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20
Weight [Mean (Standard Deviation); unit: kg] | 90 (19) | 83 (22) | 87 (21)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27 (7) | 30 (6) | 28 (7)
Fractured ribs (total) [Mean (Standard Deviation); unit: number of ribs] | 4.1 (1.4) | 3.9 (1.5) | 4.0 (1.4)
Fractured ribs (left) [Mean (Standard Deviation); unit: number of ribs] | 1.7 (1.8) | 2.0 (2.5) | 1.8 (2.1)
Fractured ribs (right) [Mean (Standard Deviation); unit: number of ribs] | 2.4 (2.3) | 1.9 (2.1) | 2.1 (2.2)
Unilateral fracture(s) [Count of Participants; unit: Participants] | 9 | 9 | 18
Bilateral fracture(s) [Count of Participants; unit: Participants] | 2 | 0 | 2
Inspiratory volume at baseline [Mean (Standard Deviation); unit: mL] | 1222 (551) | 1023 (564) | 1127 (557)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Inspired Volume
Description: maximum inspired volume measured on a handheld incentive spirometer based on the American Association of Respiratory Care (AARC) clinical practice guideline.[Restrepo. Respirated Care 2011] The best of three measurements will be recorded as the maximum inspired volume.
Time Frame: Day 1 of study treatment
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
mL | 2250 [1500 to 2500] | 1300 [750 to 2500]

2. Secondary Outcome: Maximum Inspired Volume
Description: as for outcome 1
Time Frame: Days 0, 1, 2, 7, 14, and Months 1, 1.5, and 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
mL
  Prior to intervention (baseline) | 1000 [625 to 1125] | 1000 [750 to 1500]
  Immediately following intervention | 2000 [2000 to 2625] | 1750 [1000 to 2250]
  Day 1 | 2250 [1500 to 2500] | 1300 [750 to 2500]
  Day 2 | 2250 [1500 to 2500] | 1000 [500 to 2500]
  Day 7 | 2000 [1875 to 2275] | 1750 [1225 to 3000]
  Day 14 | 2250 [2000 to 2550] | 2000 [1500 to 2775]
  Month 1 | 2500 [2200 to 2750] | 2250 [1500 to 3125]
  Month 1.5 | 2500 [2250 to 3325] | 2700 [2500 to 3375]
  Month 2 | 3000 [2500 to 3300] | 3250 [2875 to 3625]

3. Secondary Outcome: Spirometry Pain
Description: Worst pain level during the same-day spirometry use as measured using the 11-point Numeric Rating Scale with 0= no pain and 10= worst imaginable pain.
Time Frame: Days 0, 1, 2, 7, 14, and Months 1, 1.5, and 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
score on a scale
  Prior to intervention (baseline) | 10 [7 to 10] | 10 [7 to 10]
  Immediately following intervention | 3 [0 to 5] | 5 [2 to 6]
  Day 1 | 2 [0 to 7] | 8 [5 to 10]
  Day 2 | 3 [1.5 to 7] | 7 [3 to 10]
  Day 7 | 2 [0.8 to 4.8] | 7.5 [2.3 to 10]
  Day 14 | 1 [0 to 4] | 4.5 [2.8 to 6.3]
  Month 1 | 0 [0 to 2.8] | 6 [3 to 9]
  Month 1.5 | 0 [0 to 0] | 3 [1 to 9]
  Month 2 | 0 [0 to 0] | 3.8 [.8 to 7.3]

4. Secondary Outcome: Brief Pain Inventory (Pain Scale)
Description: The Brief Pain Inventory (Pain Scale) measures pain intensities: (1) worst pain; (2) least pain; (3) average pain; and (4) current pain. Each of these is measured using a 0-10 numeric rating scale, in which 0 is equivalent to no pain and 10 the worst imaginable. Then, all 4 are added together to produce a scale with values ranging from 0-40, with 0 equivalent to no pain and 40 the maximum pain.
Time Frame: Days 1, 2, and 7
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
score on a scale
  Day 1 | 7 [5 to 12] | 28 [13 to 29]
  Day 2 | 7 [6 to 12] | 21 [14 to 31]
  Day 7 | 6 [3 to 11] | 26 [16 to 31]

5. Secondary Outcome: Brief Pain Inventory (Interference Scale)
Description: The Brief Pain Inventory (Interference Scale) assesses pain's interference with physical and emotional functioning (time frame: previous 24 h). The instrument measures interference with physical and emotional functioning using a 0-10 scale (0 = no interference; 10 = complete interference). The seven interference questions involve general activity, mood, walking ability, normal work activities (both inside and outside of the home), relationships, sleep, and enjoyment of life. These seven responses are then combined to produce an interference scale (0-70), with 0 equivalent to no interference (good) and 70 equivalent to the maximum interference (bad).
Time Frame: Day 14, and Months 1, 1.5, 2, 3, 6, and 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
score on a scale
  Day 14 | 0 [0 to 16] | 30 [7 to 54]
  Month 1 | 0 [0 to 3] | 24 [6 to 58]
  Month 1.5 | 0 [0 to 0] | 1 [0 to 29]
  Month 2 | 0 [0 to 0] | 4 [0 to 11]
  Month 3 | 0 [0 to 0] | 0 [0 to 1]
  Month 6 | 0 [0 to 0] | 0 [0 to 0]
  Month 12 | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Sleep Disturbances Due to Pain
Description: Recorded as the number of awakenings subject-identified as due to pain during the previous evening
Time Frame: Days 1, 2, 7, 14; Months 1, 1.5, 2, 3, 6, and 12
Measure: Median (Inter-Quartile Range); unit: number of awakenings
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
number of awakenings
  Day 1 | 0 [0 to 1] | 2 [0 to 4]
  Day 2 | 0 [0 to 1] | 3 [1 to 5]
  Day 7 | 0 [0 to 1] | 4 [2 to 9]
  Day 14 | 0 [0 to 0] | 2 [1 to 4]
  Month 1 | 0 [0 to 0] | 1 [0 to 1]
  Month 1.5 | 0 [0 to 0] | 1 [0 to 1]
  Month 2 | 0 [0 to 0] | 0 [0 to 1]
  Month 3 | 0 [0 to 0] | 0 [0 to 1]
  Month 6 | 0 [0 to 0] | 0 [0 to 0]
  Month 12 | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Oral Opioid Consumption
Description: Recorded as the amount of oral oxycodone-equivalent analgesics consumed in previous 24 hours (measured in mg)
Time Frame: Days 1, 2, 7, 14; Months 1, 1.5, 2, 3, 6, and 12
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
mg
  Day 1 | 0 [0 to 8] | 35 [21 to 55]
  Day 2 | 0 [0 to 5] | 18 [10 to 30]
  Day 7 | 0 [0 to 2] | 15 [10 to 23]
  Day 14 | 0 [0 to 0] | 0 [0 to 6]
  Month 1 | 0 [0 to 0] | 0 [0 to 0]
  Month 1.5 | 0 [0 to 0] | 0 [0 to 1]
  Month 2 | 0 [0 to 0] | 0 [0 to 0]
  Month 3 | 0 [0 to 0] | 0 [0 to 0]
  Month 6 | 0 [0 to 0] | 0 [0 to 0]
  Month 12 | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Intravenous Opioid Consumption
Description: Recorded as the amount of intravenous morphine-equivalent analgesics consumed in previous 24 hours (measured in mg)
Time Frame: Days 1, 2, 7, 14
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
mg
  Day 1 | 0 (0) | 0 (0)
  Day 2 | 0 (0) | 0 (0)
  Day 7 | 0 (0) | 0 (0)
  Day 14 | 0 (0) | 0 (0)

9. Secondary Outcome: Day of Discharge
Description: The number of days following the study procedure of primary discharge from the hospital
Time Frame: through study completion, an average of 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
Number analyzed (Participants) | 11 | 9
days | 0.7 (1.0) | 1.4 (1.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cryoneurolysis and Placebo Intercostal Nerve Block | Sham Cryoneurolysis and Active Intercostal Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT04198662/Prot_SAP_000.pdf